CLINICAL TRIAL: NCT01527942
Title: Effect of Intravenous Acetaminophen on Postoperative Pain of Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery: A Randomized, Placebo-Controlled Trial
Brief Title: Intravenous Acetaminophen Use With Bariatric Surgery on Morbidly Obese Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Terminated per Principal Investigator's request
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 12-01-003
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2014-03

CONDITIONS: Obesity; Pain
Keywords: Pain Management
MeSH Terms: conditions — Obesity; Pain; Agnosia | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - Active Drug (Experimental): Preoperative administration of 1,000 mg IV Acetaminophen will be administered after induction of general anesthesia and prior to incision and every 6 hours thereafter for 24 hours.
  Interventions: Drug: Acetaminophen
- Arm 2 - Placebo (Placebo Comparator): Preoperative IV Placebo (0.9 Sodium Chloride 100 ml) will be administered after induction of general anesthesia and prior to incision and every 6 hours thereafter for 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Intravenous Acetaminophen 1,000 mg IV
  Other Names: OFIRMEV
  Arms: Arm 1 - Active Drug
Drug: Placebo — Placebo - IV administration 0.9% 100 ml Sodium Chloride (NaCl)
  Arms: Arm 2 - Placebo

SUMMARY:
Bariatric patients usually require the use of either intravenous or oral opioid medications. The use of opioids, however, is often associated with side-effects such as nausea, sedation pruritus, urinary retention and respiratory depression with often delay patient discharge. This study makes use of intravenous acetaminophen , a non-opioid analgesic preoperatively to determine if this will decrease the use of opioids post-operatively for pain management in morbidly obese patients undergoing laparoscopic bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly Obese and body mass index (BMI) of 35
* Between ages 20-17
* Candidates for Laparoscopic Bariatric Surgery

Exclusion Criteria:

* know hypersensitivity to acetaminophen or opioids
* impairment in liver function
* renal dysfunction
* mental retardation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Raftopoulos, MD, Principal Investigator — Saint Francis
Locations (1):
- Saint Francis Hospital, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2 - Placebo: Preoperative IV Placebo (0.9 NaCl 100 ml) will be administered after induction of general anesthesia and prior to incision and every 6 hours thereafter for 24 hours.
  Placebo: Placebo - IV administration 0.9% 100 ml NaCl
Period: Overall Study
Arm/Group | Arm 1 - Active Drug | Arm 2 - Placebo
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Active Drug | Arm 2 - Placebo | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Customized [Number; unit: Participants]
  20 to 70 Years | 16 | 18 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Relief Score on the 5-point Pain Relief Score Between Baseline and 24 Hours
Description: The 5-point Pain Relief Score is self-reported and scores range from 0=none, 1=little, 2=some, 3=a lot, 4=complete. Change = (24 hour score - baseline)
Time Frame: baseline and 24 hours
Population: Study was terminated - data were determined to be unusable by IRB due to consent issues.
Arm/Group | Arm 1 - Active Drug | Arm 2 - Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Pain Intensity on the 10-point Pain Intensity Scale Between Baseline and 24 Hours
Description: The 10-point Pain Intensity Scale is self-reported and scores range from 0=no pain to10=worst possible. Change = (24 hour score - baseline)
Time Frame: baseline and 24 hours
Population: Study was terminated - data were determined to be unusable by IRB due to consent issues.
Arm/Group | Arm 1 - Active Drug | Arm 2 - Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Response Rate - of 3=Excellent at Hour 24 Using 4-point Global Satisfaction With Regards to Overall Pain Management Rating Scale 0=Poor to 3= Excellent.
Description: The 4-point patient global satisfaction of pain management scale is self-reported and scores range from 0=poor to 3=excellent. Response rate of 3=excellent at 24 hours after baseline.
Time Frame: 24 hours after baseline
Population: Study was terminated - data were determined to be unusable by IRB due to consent issues.
Arm/Group | Arm 1 - Active Drug | Arm 2 - Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 24 hours after patients received either active drug or placebo
Arm/Group | Arm 1 - Active Drug | Arm 2 - Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Active Drug (N=16) | Arm 2 - Placebo (N=18)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Investigator determined death not related to study drug; cause of death cardiomyopathy; death occurred (4 days) outside of reporting window as defined by study protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes